CLINICAL TRIAL: NCT01099397
Title: Antihypertensive Medication Exposure as Risk for Impaired Glucose Tolerance: A PEAR Sub-Study
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: UFIRB2372009 - N; U01GM074492 (NIH)
Record Dates: First submitted 2010-04-01; First posted 2010-04-07 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Prediabetic State
Keywords: Glucose; Glucose Tolerance Test; Insulin Resistance; Metabolic adverse effects; Hypertension; Beta-blocker; Atenolol; Diuretic; Hydrochlorothiazide; Blood pressure
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Hypertension | interventions — Glucose Tolerance Test; Glucola; Sugar-Sweetened Beverages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PEAR Participants: All participants eligible for PEAR study. Each participant will be have fasting and oral glucose tolerance test data collected.
  Interventions: Other: Oral glucose tolerance test

INTERVENTIONS:
Other: Oral glucose tolerance test — For assessment of dysglycemia, 75 grams of glucose solution by mouth at 3 PEAR study visits for all enrolled participants: baseline, single drug therapy assessment, and dual drug therapy assessment.
  Other Names: OGTT; Glucose tolerance diagnostic test; Glucose tolerance test; Glucola; Sugar beverage

SUMMARY:
The purpose of this study is to determine if, in a subset of patients treated with a beta-blocker and diuretic, prediabetes is detectable to a greater extent through a 2-hour oral glucose tolerance test (OGTT) compared to fasting glucose measurement.

DETAILED DESCRIPTION:
Beta-blockers and diuretics have a well-established role in treating hypertension and are frequently used first-line. However, it is increasingly evident that these medications have harmful metabolic effects. The Pharmacogenomic Evaluation of Antihypertensive Responses (PEAR - NCT00246519) study was a greater than 700 participant, randomized, parallel assignment trial, aimed at determining the genetic factors that influence response to both a beta-blocker (atenolol) and a diuretic (hydrochlorothiazide [HCTZ]). The PEAR trial design includes evaluation at baseline, after monotherapy with either medication, and after combination therapy with both medications. This pilot, PEAR sub-study aims to characterize the ability of two diagnostics tests (fasting glucose versus glucose 2-hours after an OGTT) to detect prediabetes development prior to blood pressure medication use, after monotherapy (with atenolol or HCTZ) and after combination therapy (with atenolol and HCTZ).

ELIGIBILITY:
Inclusion Criteria:

* participation in PEAR:

  * an average seated home DBP > 85 mmHg and home SBP < 180 mmHg.
  * subjects must also have an average seated (> 5 minutes) clinic DBP between 90 mmHg and 110 mmHg and SBP < 180 mmHg.

Exclusion Criteria:

* secondary forms of HTN,
* patients currently treated with three or more antihypertensive drugs, isolated systolic HTN,
* other diseases requiring treatment with BP lowering medications,
* heart rate < 55 beats/min,
* known cardiovascular disease (including history of angina pectoris, heart failure, presence of a cardiac pacemaker, history of myocardial infarction or revascularization procedure, or cerebrovascular disease, including stroke and TIA),
* diabetes mellitus (Type 1 or 2),
* renal insufficiency (serum creatinine > 1.5 in men or 1.4 in women),
* primary renal disease,
* pregnancy or lactation,
* liver enzymes > 2.5 upper limits of normal,
* current treatment with NSAIDS,
* COX2-inhibitors,
* oral contraceptives or estrogen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic, PEAR participants
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Johnson, PharmD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Department of Community Health and Family Medicine, Gainesville, Florida, United States

REFERENCES:
- See also: Pharmacogenomic Evaluation of Antihypertensive Responses (PEAR) ClinicalTrials website — http://clinicaltrials.gov/ct2/show/NCT00246519?term=NCT00246519&rank=1

RESULTS

PARTICIPANT FLOW:
Groups:
- PEAR Sub-study Participants: All participants eligible for the PEAR study in Gainesville, FL, starting May 2009, were allowed to participate in the PEAR sub-study; participants enrolled were evaluated at three time points as part of the PEAR protocol, at baseline, 9 weeks and 18 weeks; for each participant at each time point, a fasting glucose value and 2-hour oral glucose tolerance test value was collected and compared
Period: Overall Study
Arm/Group | PEAR Sub-study Participants
Started | 39
Completed | 26
Not Completed | 13
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Groups:
- PEAR Sub-study Participants: All participants eligible for the PEAR study in Gainesville, FL, starting May 2009, were allowed to participate in the PEAR sub-study
Arm/Group | PEAR Sub-study Participants
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Diagnosed With Prediabetes or Normal Glucose, by 2 Measurements (Fasting Glucose Measurement and Glucose Measurement After a 2-hour Oral Glucose Tolerance Test [OGTT]), at Three Timepoints During Antihypertensive Treatment
Description: A single cohort of patients was followed through participation in the parent study, PEAR, and had both fasting and 2-hour OGTT labs evaluated at three time points. At each of these time points the two methods for evaluating prediabetes were compared. Consistent with the definition for prediabetes recommended by the American Diabetes Association, a fasting glucose above 99mg/dL or 2-hour oral glucose tolerance test glucose above 139mg/dL was considered prediabetic for this study.
Time Frame: Baseline, 9 weeks, and 18 weeks after initiation of PEAR intervention(s)
Population: Only including participants with data at each time point
Measure: Number; unit: participants
Groups:
- 2-hour Glucose: Glucose collected after a 2 hour oral glucose tolerance test
- Fasting Glucose: Fasting glucose collected
Arm/Group | 2-hour Glucose | Fasting Glucose
Number analyzed (Participants) | 26 | 26
participants
  Prediabetic at baseline | 6 | 8
  Normal glucose at baseline | 20 | 18
  Prediabetic at 9 weeks | 7 | 9
  Normal glucose at 9 weeks | 19 | 17
  Prediabetic at 18 weeks | 7 | 9
  Normal glucose at18 weeks | 15 | 13
Statistical Analysis 1: Comparison: 2-hour Glucose vs Fasting Glucose; p<0.05 was considered significant at baseline; the null hypothesis was that there was no difference between prediabetes diagnosis (by 2-hour glucose or fasting glucose), the alternative hypothesis was that there was a significant difference between prediabetes diagnosis (by 2-hour glucose or fasting glucose); Test type: Superiority or Other; p = 0.41, McNemar — P-value at baseline; McNemar was used at each of three time points to compare prediabetes diagnosis by fasting versus 2-hour OGTT
Statistical Analysis 2: Comparison: 2-hour Glucose vs Fasting Glucose; p<0.05 was considered significant at 9 week assessment; the null hypothesis was that there was no difference between prediabetes diagnosis (by 2-hour glucose or fasting glucose), the alternative hypothesis was that there was a significant difference between prediabetes diagnosis (by 2-hour glucose or fasting glucose); Test type: Superiority or Other; p = 0.59, McNemar — P-value at 9 weeks; McNemar was used at each of three time points to compare prediabetes diagnosis by fasting versus 2-hour OGTT
Statistical Analysis 3: Comparison: 2-hour Glucose vs Fasting Glucose; p<0.05 was considered significant at 18 week assessment; the null hypothesis was that there was no difference between prediabetes diagnosis (by 2-hour glucose or fasting glucose), the alternative hypothesis was that there was a significant difference between prediabetes diagnosis (by 2-hour glucose or fasting glucose); Test type: Superiority or Other; p = 0.41, McNemar — P-value at 18 weeks; McNemar was used at each of three time points to compare prediabetes diagnosis by fasting versus 2-hour OGTT

ADVERSE EVENTS:
Groups:
- PEAR Sub-study Participants: All participants in the PEAR sub-study were evaluated by two methods at 3 time-points in the PEAR parent study
Arm/Group | PEAR Sub-study Participants
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

LIMITATIONS AND CAVEATS:
This was a pilot study to evaluate two glucose phenotypes in a small sample from a larger trial. As such, our sample size was small. Further, if participants were withdrawn from the parent trial, they were also withdrawn from the sub-study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes